CLINICAL TRIAL: NCT00878189
Title: A PHASE I TRIAL OF PF-03084014 IN PATIENTS WITH ADVANCED SOLID TUMOR MALIGNANCY AND T-CELL ACUTE LYMPHOBLASTIC LEUKEMIA/LYMPHOBLASTIC LYMPHOMA
Brief Title: A Trial In Patients With Advanced Cancer And Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A8641014; 2010-022036-36 (EudraCT Number)
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Neoplasms by Histologic Type
Keywords: Phase 1 dose escalation study in advanced solid tumor malignancy and leukemia
MeSH Terms: conditions — Neoplasms by Histologic Type; Leukemia | interventions — nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-03084014

INTERVENTIONS:
Drug: PF-03084014 — 10 mg, 50 mg or 100 mg tablets. Patients dosed from 20 mg - 500 mg, twice daily
  Other Names: gamma secretase inhibitor

SUMMARY:
This is a phase 1, dose escalating study to determine the safety of PF-03084014 in patients with advanced cancer and leukemia

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced cancer that is resistant to standard therapy or for which no standard therapy is available
* Patients with acute T cell leukemia/lymphoblastic lymphoma that is resistant to standard therapy or for which no standard therapy is available
* Men and women >16 years old

Exclusion Criteria:

* Prior treatment with a gamma secretase inhibitor for treatment of cancer
* Patients taking Tamoxifen
* Patients with active graft versus host disease
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
* Patients who are pregnant or breast feeding
* Patients with clinical evidence of central nervous system disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-06-25 (Actual); Primary Completion 2013-01-10 (Actual); Study Completion 2016-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (8):
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Denver CTRC, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Massachusetts General Hospital Clinical Laboratory, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Ferber Cancer institute, Boston, Massachusetts
  - Karmanos Cancer Center / Wayne State University, Detroit, Michigan
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Italy (2):
  - DIPRTMNT CLIN Scienze RADIOL e Istocitopatologiche, Bologna
  - Istituto di Ematologia Seragnoli, Bologna

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Papayannidis C, DeAngelo DJ, Stock W, Huang B, Shaik MN, Cesari R, Zheng X, Reynolds JM, English PA, Ozeck M, Aster JC, Kuo F, Huang D, Lira PD, McLachlan KR, Kern KA, Garcia-Manero G, Martinelli G. A Phase 1 study of the novel gamma-secretase inhibitor PF-03084014 in patients with T-cell acute lymphoblastic leukemia and T-cell lymphoblastic lymphoma. Blood Cancer J. 2015 Sep 25;5(9):e350. doi: 10.1038/bcj.2015.80. No abstract available. PMID 26407235
- [Derived] Tabares-Seisdedos R, Rubenstein JL. Inverse cancer comorbidity: a serendipitous opportunity to gain insight into CNS disorders. Nat Rev Neurosci. 2013 Apr;14(4):293-304. doi: 10.1038/nrn3464. PMID 23511909
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8641014&StudyName=A%20Trial%20In%20Patients%20With%20Advanced%20Cancer%20And%20Leukemia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study originally planned to give PF-03084014 in combination with dexamethasone in participants with solid tumors and with T-cell acute lymphoblastic leukemia and lymphoblastic lymphoma, including a drug-drug-interaction test of PF-03084014 and dexamethasone in solid tumor participants. But these parts were removed per protocol amendments.
Groups:
- PF-03084014 20 mg BID in Solid Tumor Participants: PF-03084014 20 mg was administered orally twice daily (BID), beginning on Day 1 of each cycle, for 21 days. In Cycle 1 only, participants with advanced solid tumor malignancies received PF-03084014 BID for 21 days (on Cycle 1 Day 21 only the morning dose was administered) followed by 7 days' off-treatment for the purpose of pharmacokinetic (PK) assessments. In Cycle 2 and beyond, PF-03084014 was administered BID continuously.
- PF-03084014 40 mg BID in Solid Tumor Participants: PF-03084014 40 mg was administered orally BID, beginning on Day 1 of each cycle, for 21 days. In Cycle 1 only, participants with advanced solid tumor malignancies received PF-03084014 BID for 21 days (on Cycle 1 Day 21 only the morning dose was administered) followed by 7 days' off-treatment for the purpose of PK assessments. In Cycle 2 and beyond, PF-03084014 was administered BID continuously.
- PF-03084014 80 mg BID in Solid Tumor Participants: PF-03084014 80 mg was administered orally BID, beginning on Day 1 of each cycle, for 21 days. In Cycle 1 only, participants with advanced solid tumor malignancies received PF-03084014 BID for 21 days (on Cycle 1 Day 21 only the morning dose was administered) followed by 7 days' off-treatment for the purpose of PK assessments. In Cycle 2 and beyond, PF-03084014 was administered BID continuously.
- PF-03084014 100 mg BID in Solid Tumor Participants: PF-03084014 100 mg was administered orally BID, beginning on Day 1 of each cycle, for 21 days. In Cycle 1 only, participants with advanced solid tumor malignancies received PF-03084014 BID for 21 days (on Cycle 1 Day 21 only the morning dose was administered) followed by 7 days' off-treatment for the purpose of PK assessments. In Cycle 2 and beyond, PF-03084014 was administered BID continuously.
- PF-03084014 130 mg BID in Solid Tumor Participants: PF-03084014 130 mg was administered orally BID, beginning on Day 1 of each cycle, for 21 days. In Cycle 1 only, participants with advanced solid tumor malignancies received PF-03084014 BID for 21 days (on Cycle 1 Day 21 only the morning dose was administered) followed by 7 days' off-treatment for the purpose of PK assessments. In Cycle 2 and beyond, PF-03084014 was administered BID continuously.
- PF-03084014 150 mg BID in Solid Tumor Participants: PF-03084014 150 mg was administered orally BID, beginning on Day 1 of each cycle, for 21 days. In Cycle 1 only, participants with advanced solid tumor malignancies received PF-03084014 BID for 21 days (on Cycle 1 Day 21 only the morning dose was administered) followed by 7 days' off-treatment for the purpose of PK assessments. In Cycle 2 and beyond, PF-03084014 was administered BID continuously.
- PF-03084014 220 mg BID in Solid Tumor Participants: PF-03084014 220 mg was administered orally BID, beginning on Day 1 of each cycle, for 21 days. In Cycle 1 only, participants with advanced solid tumor malignancies received PF-03084014 BID for 21 days (on Cycle 1 Day 21 only the morning dose was administered) followed by 7 days' off-treatment for the purpose of PK assessments. In Cycle 2 and beyond, PF-03084014 was administered BID continuously.
- PF-03084014 330 mg BID in Solid Tumor Participants: PF-03084014 330 mg was administered orally BID, beginning on Day 1 of each cycle, for 21 days. In Cycle 1 only, participants with advanced solid tumor malignancies received PF-03084014 BID for 21 days (on Cycle 1 Day 21 only the morning dose was administered) followed by 7 days' off-treatment for the purpose of PK assessments. In Cycle 2 and beyond, PF-03084014 was administered BID continuously.
- PF-03084014 150 mg BID in T-ALL/LBL Participants: PF-03084014 150 mg was administered orally BID to participants with T-cell acute lymphoblastic leukemia/lymphoblastic lymphoma (T-ALL/LBL) as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
Period: Overall Study
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Started | 3 | 3 | 4 | 8 | 4 | 23 | 16 | 3 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 8 | 4 | 23 | 16 | 3 | 8
Not completed — Death | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Participant Refused to Follow-up | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Other | 3 | 2 | 4 | 7 | 4 | 18 | 15 | 3 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Objection Progression or Relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- PF-03084014 in Solid Tumor Participants: PF-03084014 was administered orally BID, beginning on Day 1 of each cycle, for 21 days. In Cycle 1 only, participants with advanced solid tumor malignancies received PF-03084014 BID for 21 days (on Cycle 1 Day 21 only the morning dose was administered) followed by 7 days' off-treatment for the purpose of PK assessments. In Cycle 2 and beyond, PF-03084014 was administered BID continuously.
- PF-03084014 in T-ALL/LBL Participants: PF-03084014 150 mg was administered orally BID to participants with T-ALL/LBL as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
- Total: Total of all reporting groups
Arm/Group | PF-03084014 in Solid Tumor Participants | PF-03084014 in T-ALL/LBL Participants | Total
Number analyzed (Participants) | 64 | 8 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (14.7) | 30.8 (9) | 52.9 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 2 | 35
  Male | 31 | 6 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Solid Tumor Participants With First-Cycle Dose-Limiting Toxicity (DLT)
Description: Any DLT event attributable to PF-03084014 during Cycle 1: non-hematologic toxicities >= Grade 3 despite optimal care; treatment delay >=7 days or unable to deliver at least 80% of planned dose due to treatment-related toxicities; Grade 4 neutropenia >7 days; febrile neutropenia; neutropenic infection; Grade >=3 thrombocytopenia with bleeding
Time Frame: Baseline to the end of Cycle 1 (Week 4)
Population: Solid tumor participants enrolled for dose-escalation who started treatment and who did not have first cycle major treatment deviations (including less than 80% of the planned dose of PF-03084014 in Cycle 1 for reasons other than treatment-related toxicities) were evaluable for DLTs.
Measure: Number; unit: participants
Groups:
- PF-03084014 20 mg BID in Solid Tumor Participants: PF-03084014 20 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
- PF-03084014 40 mg BID in Solid Tumor Participants: PF-03084014 40 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
- PF-03084014 80 mg BID in Solid Tumor Participants: PF-03084014 80 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
- PF-03084014 100 mg BID in Solid Tumor Participants: PF-03084014 100 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
- PF-03084014 130 mg BID in Solid Tumor Participants: PF-03084014 130 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
- PF-03084014 150 mg BID in Solid Tumor Participants: PF-03084014 150 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
- PF-03084014 220 mg BID in Solid Tumor Participants: PF-03084014 220 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
- PF-03084014 330 mg BID in Solid Tumor Participants: PF-03084014 330 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 6 | 6 | 2
participants | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2

2. Primary Outcome: Number of T-ALL/LBL Participants With First-Cycle DLT
Description: Any DLT attributable to PF-03084014 at 1st Cycle: non-hematologic toxicities >= Grade 3 despite optimal care; treatment delay >=7 days; unable to deliver at least 80% of planned dose; absolute neutrophil count (ANC) <1000/microliter (uL), or platelet count <30,000/uL, or hemoglobin <8 gram/deciliter (g/dL) in a bone marrow with <5% blasts and no evidence of leukemia or abnormal dysplasia for >42 days
Time Frame: Baseline to the end of Cycle 1 (Week 4)
Population: T-ALL/LBL participants enrolled for dose-escalation who started treatment and who did not have first cycle major treatment deviations (including less than 80% of the planned dose of PF-03084014 in Cycle 1 for reasons other than treatment-related toxicities) were evaluable for DLTs.
Measure: Number; unit: participants
Arm/Group | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 5
participants | 1

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) (All Causality)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of casual relationship. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death, was life-threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), and resulted in congenital anomaly/birth defect.
Time Frame: Baseline up to end of study (maximum of 84 months)
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- PF-03084014 20 mg BID in Solid Tumor Participants: PF-03084014 20 mg was administered orally twice daily (BID) to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 4 | 23 | 16 | 3 | 8
participants
  No. of Participants With AEs | 3 | 3 | 4 | 7 | 4 | 23 | 16 | 3 | 8
  No. of Participants With SAEs | 1 | 1 | 2 | 4 | 2 | 8 | 7 | 2 | 4
  No. of Participants Discontinued PF-03084014 | 0 | 1 | 0 | 2 | 1 | 1 | 4 | 2 | 3
  No. of Participants Temp. Discontinued Treatment | 1 | 1 | 2 | 1 | 1 | 9 | 5 | 1 | 0
  No. of Participants With Dose Reduction Due to AEs | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 1 | 1

4. Secondary Outcome: Number of Participants With TEAEs (Treatment-Related)
Description: An AE was any untoward medical occurrence in a participant who received study drug. Treatment-related events were those assessed by the investigator as related to study medication. An SAE was any untoward medical occurrence at any dose that: resulted in death, was life-threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), and resulted in congenital anomaly/birth defect.
Time Frame: Baseline up to end of study (maximum of 84 months)
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 4 | 23 | 16 | 3 | 8
participants
  No. of Participants With AEs | 2 | 1 | 2 | 6 | 4 | 20 | 16 | 3 | 5
  No. of Participants With SAEs | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
  No. of Participants Discontinued PF-03084014 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  No. of Participants Temp. Discontinued Treatment | 0 | 0 | 0 | 0 | 1 | 7 | 4 | 1 | 0
  No.of Participants With Dose Reduction Due to AEs | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 1 | 1

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) (All Causality) by Severity (by Maximum Common Terminology Criteria for Adverse Events [CTCAE] Grade)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. CTCAE version 3.0 was used for AE grading: Grade 1 mild AE; Grade 2 moderate AE; Grade 3 severe AE; Grade 4 life-threatening or disabling AE; Grade 5 death related to AE.
Time Frame: Baseline up to end of study (maximum of 84 months)
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 4 | 23 | 16 | 3 | 8
participants
  Any AEs, Grade 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1
  Any AEs, Grade 2 | 2 | 1 | 0 | 1 | 2 | 8 | 3 | 0 | 1
  Any AEs, Grade 3 | 1 | 1 | 2 | 2 | 2 | 12 | 9 | 2 | 4
  Any AEs, Grade 4 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 1 | 1
  Any AEs, Grade 5 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1

6. Secondary Outcome: Number of Participants With TEAEs (Treatment-Related) by Severity (by Maximum CTCAE Grade)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-related events were those assessed by the investigator as related to study medication. CTCAE version 3.0 was used for AE grading: Grade 1 mild AE; Grade 2 moderate AE; Grade 3 severe AE; Grade 4 life-threatening or disabling AE; Grade 5 death related to AE.
Time Frame: Baseline up to end of study (maximum of 84 months)
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 4 | 23 | 16 | 3 | 8
participants
  Any AEs, Grade 1 | 1 | 0 | 1 | 1 | 1 | 6 | 2 | 0 | 3
  Any AEs, Grade 2 | 1 | 1 | 0 | 3 | 2 | 6 | 4 | 1 | 0
  Any AEs, Grade 3 | 0 | 0 | 1 | 1 | 1 | 8 | 10 | 2 | 1
  Any AEs, Grade 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Any AEs, Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing or Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

7. Secondary Outcome: Number of Participants With Potentially Clinical Significant Categorical Changes From Baseline in Electrocardiogram (ECG) Findings in QTc Interval
Description: Criteria for potentially important changes in ECG were defined as: maximum (max.) post-dose (post-baseline) time from electrocardiogram Q wave to the corresponding to electrical systole (QT interval) corrected for Fridericia's factor (QTcF), or QT interval corrected for Bazett's factor (QTcB): <450, 450 -<480, 480-<500, and >=500 msec. Maximum increase (inc.) from baseline in QTcF or QTcB: change (chg) <30, 30>=chg<60, and chg >=60 msec.
Time Frame: Baseline up to end of study (maximum of 84 months)
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 4 | 23 | 16 | 3 | 8
participants
  Max. QTcB interval <450 msec | 0 | 3 | 2 | 4 | 2 | 11 | 5 | 2 | 8
  Max. QTcB interval 450-<480 msec | 3 | 0 | 1 | 3 | 2 | 8 | 9 | 1 | 8
  Max. QTcB interval 480-<500 msec | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 8
  Max. QTcB interval >=500 msec | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 8
  Max. QTcF interval <450 msec | 3 | 3 | 2 | 7 | 3 | 13 | 12 | 3 | 8
  Max. QTcF interval 450-<480 msec | 0 | 0 | 1 | 0 | 1 | 9 | 2 | 0 | 0
  Max. QTcF interval 480-<500 msec | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Max. QTcF interval >=500 msec | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
  Max. QTcB interval inc. from baseline chg<30 msec | 1 | 2 | 1 | 7 | 3 | 21 | 7 | 3 | 7
  Max. QTcB interval inc. from baseline 30=<chg<60 | 2 | 1 | 2 | 1 | 1 | 2 | 7 | 0 | 1
  Max. QTcB interval inc. from baseline chg>=60 msec | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
  Max. QTcF interval inc. from baseline chg<30 msec | 3 | 2 | 1 | 7 | 3 | 22 | 12 | 3 | 8
  Max. QTcF interval inc. from baseline 30=<chg<60 | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 0 | 0
  Max. QTcF interval inc. from baseline chg>=60 msec | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0

8. Secondary Outcome: Number of Participants With Laboratory Tests Abnormalities Meeting the Criteria of Potential Clinical Concern (Hematology and Chemistries, All Cycles)
Description: Parameters analyzed included: white blood cell (WBC) count plus differential, absolute (abs) neutrophil count, platelets, hemoglobin, sodium, potassium, bicarbonate, chloride, blood urea nitrogen, creatinine, glucose, uric acid, calcium, phosphate, magnesium, total protein, albumin, total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), partial prothrombin time/international normalized ratio (PTT/INR). Urinalysis: pH, specific gravity, protein, glucose, ketones, blood, leukocyte esterase, and nitrites. Pregnancy test: Serum or urine pregnancy test for women of childbearing potential. There were no changes in urine protein among the solid tumor and T-ALL/LBL participants that were clinically significant. Clinical significance was judged by the investigator.
Time Frame: Baseline up to end of study (maximum of 84 months)
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- PF-03084014 in Solid Tumor Participants: PF-03084014 20, 40, 80, 100, 150, 220, 330 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
Arm/Group | PF-03084014 in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 64 | 8
participants
  Hemoglobin | 45 | 8
  Lymphocytes (abs) | 40 | 8
  Neutrophils (abs) | 4 | 5
  Platelets | 13 | 6
  WBC | 4 | 5
  ALT | 22 | 4
  ALP | 24 | 3
  AST | 32 | 4
  Bicarbonate | 15 | 1
  Bilirubin | 10 | 2
  Creatinine | 17 | 1
  Hypercalcaemia | 17 | 0
  Hyperglycaemia | 55 | 6
  Hyperkalaemia | 4 | 0
  Hypermagnesaemia | 1 | 0
  Hypernatraemia | 4 | 0
  Hypoalbuminaemia | 43 | 6
  Hypocalcaemia | 18 | 6
  Hypoglycaemia | 6 | 0
  Hypokalaemia | 23 | 4
  Hypomagnesaemia | 8 | 1
  Hyponatraemia | 19 | 3
  Hypophosphataemia | 54 | 4

9. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) After a Single Dose on Cycle 1 Day 1
Description: Cmax was the maximum observed serum concentration.
Time Frame: Cycle 1 Day 1 (pre-dose and 0.5, 1, 2, 4, and 10 hr post-dose)
Population: All treated participants who had at least 1 of the PK parameters of interest. N=number of participants evaluable for this outcome measure (OM).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 4 | 22 | 16 | 3 | 8
nanogram/milliliter (ng/mL) | 163 (62) | 368 (48) | 230 (193) | 691 (37) | 536 (72) | 943 (100) | 861 (63) | 1892 (54) | 1604 (85)

10. Secondary Outcome: Dose-normalized Cmax [Cmax (dn)] After a Single Dose on Cycle 1 Day 1
Description: Cmax(dn) was calculated by maximum observed serum concentration (Cmax) divided by administered dose.
Time Frame: Cycle 1 Day 1 (pre-dose and 0.5, 1, 2, 4, and 10 hr post-dose)
Population: All treated participants who had at least 1 of the PK parameters of interest. N=number of participants evaluable for this OM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 4 | 22 | 16 | 3 | 8
ng/mL/mg | 8.1 (63) | 9.2 (48) | 2.9 (193) | 6.9 (37) | 4.1 (72) | 6.3 (100) | 3.9 (63) | 5.7 (54) | 10.7 (85)

11. Secondary Outcome: Area Under the Time-Concentration Curve From Time 0 to the Dosing Interval (AUCtau) After a Single Dose on Cycle 1 Day 1
Description: AUCtau was area under the serum concentration-time profile from time 0 to tau (dosing interval). CV is the coefficient of variation.
Time Frame: Cycle 1 Day 1 (pre-dose and 0.5, 1, 2, 4, and 10 hr post-dose)
Population: All treated participants who had at least 1 of the PK parameters of interest. Overall Number of Participants Analyzed (N) =number of participants evaluable for this outcome measure (OM).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 3 | 21 | 16 | 2 | 4
nanogram*hour/milliliter (ng*hr/mL) | 409 (83) | 1329 (87) | 1649 (98) | 2204 (37) | 2924 (81) | 3677 (86) | 3593 (58) | 8014 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric % CV was not calculated. | 6412 (80)

12. Secondary Outcome: Dose-normalized AUCtau [AUCtau (dn) ] After a Single Dose on Cycle 1 Day 1
Description: AUCtau (dn) was calculated by area under the serum concentration-time profile from time 0 to tau (dosing interval) (AUCtau) divided by administered dose. NE is not estimable.
Time Frame: Cycle 1 Day 1 (pre-dose and 0.5, 1, 2, 4, and 10 hr post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 3 | 21 | 16 | 2 | 4
ng*hr/mL/mg | 20.4 (83) | 33.2 (87) | 20.6 (98) | 22.0 (37) | 22.5 (81) | 24.5 (86) | 16.3 (58) | 24.3 (NA) — Geometric %CV was NE when No. of subjects analyzed is <3, hence data was not calculated. | 42.7 (80)

13. Secondary Outcome: Time to Reach Cmax (Tmax) After a Single Dose on Cycle 1 Day 1
Description: Tmax was the time to reach maximum serum concentration (Cmax).
Time Frame: Cycle 1 Day 1 (pre-dose and 0.5, 1, 2, 4, and 10 hr post-dose)
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 4 | 23 | 16 | 3 | 8
hours | 1.0 [0.9 to 1.0] | 1.0 [1.0 to 1.3] | 2.0 [1.0 to 8.0] | 1.0 [1.0 to 2.0] | 2.5 [1.0 to 4.0] | 1.1 [0.5 to 4.1] | 2.0 [1.0 to 4.1] | 1.2 [1.0 to 2.0] | 1.1 [0.9 to 4.0]

14. Secondary Outcome: Cmax After Multiple Dose on Cycle 1 Day 21
Description: Cmax was the maximum observed serum concentration. Cycle 1 Day 21 PK parameter summaries are presented only for participants who were considered to be dose compliant. CV is the coefficient of variation.
Time Frame: Cycle 1 Day 21 (pre-dose and 0.5, 1, 2, 4, 10, 24, 48, 96 and 120 hr post-dose)
Population: All participants who had at least 6 days of uninterrupted dosing prior to the Cycle 1 Day 21 PK assessment. The 6-day duration was chosen based on the observed terminal half-life of PF-03084014. N=number of participants evaluable for this OM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 2 | 2 | 3 | 5 | 3 | 12 | 8 | 4
ng/mL | 64.5 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 381 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 313 (29) | 867 (44) | 421 (130) | 1246 (79) | 1864 (76) | 1828 (42)

15. Secondary Outcome: Time to Reach Cmax (Tmax) After Multiple Dose on Cycle 1 Day 21
Description: Tmax was the time to reach maximum serum concentration (Cmax). Cycle 1 Day 21 PK parameter summaries are presented only for participants who were considered to be dose compliant.
Time Frame: Cycle 1 Day 21 (pre-dose and 0.5, 1, 2, 4, 10, 24, 48, 96 and 120 hr post-dose)
Population: as for outcome 14
Measure: Median (Full Range); unit: hour
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 2 | 2 | 3 | 5 | 3 | 12 | 8 | 4
hour | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0] | 1.1 [1.0 to 4.0] | 1.0 [1.0 to 2.7] | 3.7 [1.0 to 8.0] | 1.1 [1.0 to 4.0] | 1.0 [0.5 to 2.0] | 1.6 [1.0 to 2.0]

16. Secondary Outcome: AUCtau After Multiple Dose on Cycle 1 Day 21
Description: AUCtau was area under the serum concentration-time profile from time 0 to tau (dosing interval). Cycle 1 Day 21 PK parameter summaries are presented only for participants who were considered to be dose compliant.
Time Frame: Cycle 1 Day 21 (pre-dose and 0.5, 1, 2, 4, 10, 24, 48, 96 and 120 hr post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 2 | 2 | 3 | 5 | 3 | 12 | 8 | 4
ng*hr/mL | 309.0 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 2521 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 1572 (42) | 4741 (70) | 3155 (59) | 6430 (89) | 10520 (89) | 9161 (30)

17. Secondary Outcome: Apparent Volume of Distribution (Vz/F) on Cycle 1 Day 21
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired concentration of a drug. Cycle 1 Day 21 PK parameter summaries are presented only for participants who were considered to be dose compliant.
Time Frame: Cycle 1 Day 21 (pre-dose and 0.5, 1, 2, 4, 10, 24, 48, 96 and 120 hr post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 3 | 12 | 8 | 3
liter (L) | 2810 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 516 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 3353 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 986 (52) | 2048 (49) | 801 (144) | 852 (120) | 424 (61)

18. Secondary Outcome: Serum Decay Half-Life (t1/2) After Multiple Dose on Cycle 1 Day 21
Description: Serum decay half-life (t1/2) is the time measured for the serum concentration to decrease by one half. Cycle 1 Day 21 PK parameter summaries are presented only for participants who were considered to be dose compliant.
Time Frame: Cycle 1 Day 21 (pre-dose and 0.5, 1, 2, 4, 10, 24, 48, 96 and 120 hr post-dose)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 3 | 12 | 8 | 3
hours | 30.3 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 22.6 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated.. | 38.6 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 34.2 (11.7) | 34.7 (5.3) | 25.3 (9.2) | 29.3 (9.3) | 18.0 (3.6)

19. Secondary Outcome: Apparent Oral Clearance (CL/F) on Cycle 1 Day 21
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Cycle 1 Day 21 PK parameter summaries are presented only for participants who were considered to be dose compliant.
Time Frame: Cycle 1 Day 21 (pre-dose and 0.5, 1, 2, 4, 10, 24, 48, 96 and 120 hr post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour (L/hr)
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 2 | 2 | 3 | 5 | 3 | 12 | 8 | 4
liter/hour (L/hr) | 64.8 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 15.9 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 50.9 (42) | 21.1 (70) | 41.2 (59) | 23.4 (88) | 20.9 (89) | 16.4 (30)

20. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) After Multiple Dose on Cycle 1 Day 21
Description: Cmin was the minimum serum concentration. Cycle 1 Day 21 PK parameter summaries are presented only for participants who were considered to be dose compliant.
Time Frame: Cycle 1 Day 21 (pre-dose and 0.5, 1, 2, 4, 10, 24, 48, 96 and 120 hr post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 2 | 2 | 3 | 5 | 3 | 12 | 8 | 4
ng/mL | 10.7 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 126 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 59.2 (103) | 232 (118) | 206 (40) | 266 (102) | 469 (118) | 420 (81)

21. Secondary Outcome: Average Serum Concentration (Cavg) at Steady State on Cycle 1 Day 21
Description: Cavg was the average serum concentration at steady state. Cycle 1 Day 21 PK parameter summaries are presented only for participants who were considered to be dose compliant.
Time Frame: Cycle 1 Day 21 (pre-dose and 0.5, 1, 2, 4, 10, 24, 48, 96 and 120 hr post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 2 | 2 | 3 | 5 | 3 | 12 | 8 | 4
ng/mL | 25.7 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 210 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 131 (42) | 395 (69) | 263 (59) | 536 (89) | 877 (89) | 763 (30)

22. Secondary Outcome: Accumulation Ratio (Rac) on Cycle 1 Day 21
Description: Accumulation was calculated as AUCtau at steady state (Cycle 1 Day 21) divided by AUCtau after a single dose on Cycle 1 Day 1. Cycle 1 Day 21 PK parameter summaries are presented only for participants who were considered to be dose compliant.
Time Frame: Cycle 1 Day 1 (pre-dose and 0.5, 1, 2, 4, and 10 hr post-dose), Cycle 1 Day 21 (pre-dose and 0.5, 1, 2, 4, 10, 24, 48, 96 and 120 hr post-dose)
Population: as for outcome 14
Measure: Median (Full Range); unit: ratio
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 3 | 12 | 8 | 1
ratio | 1.18 [0.72 to 1.63] | 1.60 [1.45 to 1.74] | 1.36 [0.93 to 1.79] | 2.49 [1.23 to 2.86] | 1.98 [1.81 to 2.15] | 2.29 [0.95 to 4.90] | 2.84 [1.14 to 5.80] | 0.97 [NA to NA] — Unable to calculate as only 1 participant provided value.

23. Secondary Outcome: Dose-normalized AUCtau [AUCtau (dn)] After Multiple Dose on Cycle 1 Day 21
Description: AUCtau (dn) was calculated by area under the serum concentration-time profile from time 0 to tau (dosing interval) (AUCtau) divided by administered dose. Cycle 1 Day 21 PK parameter summaries are presented only for participants who were considered to be dose compliant.
Time Frame: Cycle 1 Day 21 (pre-dose and 0.5, 1, 2, 4, 10, 24, 48, 96 and 120 hr post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 2 | 2 | 3 | 5 | 3 | 12 | 8 | 4
ng*hr/mL/mg | 15.4 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 63.0 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 19.7 (41) | 47.4 (70) | 24.3 (59) | 42.9 (88) | 47.9 (89) | 61.1 (30)

24. Secondary Outcome: Dose-normalized Cmax [Cmax (dn)] After Multiple Dose on Cycle 1 Day 21
Description: Cmax(dn) was calculated by maximum observed serum concentration (Cmax) divided by administered dose. Cycle 1 Day 21 PK parameter summaries are presented only for participants who were considered to be dose compliant.
Time Frame: Cycle 1 Day 21 (pre-dose and 0.5, 1, 2, 4, 10, 24, 48, 96 and 120 hr post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 2 | 2 | 3 | 5 | 3 | 12 | 8 | 4
ng/mL/mg | 3.2 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 9.6 (NA) — Geometric %CV was not estimable when number of participants analyzed is less than 3, hence data for Geometric %CV was not calculated. | 3.9 (29) | 8.7 (44) | 3.2 (130) | 8.3 (79) | 8.5 (76) | 12.2 (42)

25. Secondary Outcome: AUCtau in the Fasted State for Solid Tumor Participants
Description: AUCtau was area under the serum concentration-time profile from time 0 to tau (dosing interval).
Time Frame: Cycle 1 Day 1 (pre-dose and 0.5, 1, 2, 4, 10 and 24 hr post-dose) or Cycle 2 Day 1 (pre-dose and 0.5, 1, 2, 4, 10 and 24 hr post-dose)
Population: Solid tumor participants who were enrolled in the food-effect sub-study, were treated and had evaluable PK data under both fed and fasted states.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- PF-03084014 150 mg BID in Solid Tumor Participants: PF-03084014 150 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1=28 days [with a 7-day washout]). On Cycle 1 Day 1 and Cycle 2 Day 1, only the morning dose was administered. Each participant was to serve as their own control in which PF-03084014 was administered in the morning under either "fed" or "fasted" conditions on Day 1 of Cycle 1 and Cycle 2. The testing order for fed versus fasted conditions was as follows: The first 6 participants in this sub-study were tested under fed followed by fasted conditions, the next 6 participants were tested under fasted followed by fed conditions.
- PF-03084014 220 mg BID in Solid Tumor Participants: PF-03084014 220 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1=28 days [with a 7-day washout]). On Cycle 1 Day 1 and Cycle 2 Day 1, only the morning dose was administered. Each participant was to serve as their own control in which PF-03084014 was administered in the morning under either "fed" or "fasted" conditions on Day 1 of Cycle 1 and Cycle 2. The testing order for fed versus fasted conditions was as follows: The first 6 participants in this sub-study were tested under fed followed by fasted conditions, the next 6 participants were tested under fasted followed by fed conditions.
Arm/Group | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 7 | 4
ng*hr/mL | 2547 (101) | 9353 (100)

26. Secondary Outcome: AUCtau in the Fed State for Solid Tumor Participants
Description: AUCtau was area under the serum concentration-time profile from time 0 to tau (dosing interval).
Time Frame: as for outcome 25
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 7 | 4
ng*hr/mL | 3163 (83) | 5573 (39)

27. Secondary Outcome: Cmax in the Fasted State for Solid Tumor Participants
Description: Cmax was the maximum observed serum concentration.
Time Frame: as for outcome 25
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 9 | 4
ng/mL | 795.1 (104) | 2334 (93)

28. Secondary Outcome: Cmax in the Fed State for Solid Tumor Participants
Description: Cmax was the maximum observed serum concentration.
Time Frame: as for outcome 25
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 9 | 4
ng/mL | 862.3 (74) | 924.4 (40)

29. Secondary Outcome: Dose-normalized AUCtau [AUCtau(dn)] in the Fasted State for Solid Tumor Participants
Description: AUCtau(dn) was calculated by area under the serum concentration-time profile from time 0 to tau (dosing interval) (AUCtau) divided by administered dose.
Time Frame: as for outcome 25
Population: Solid tumor participants who were enrolled in the food-effect sub-study, were treated and had evaluable PK data under both fed and fasted states. Due to the limited number of evaluable participants (7 at 150 mg BID and 4 at 220 mg BID for Cmax) and a generally dose-proportional exposure (AUCtau and Cmax), data were combined for the 2 dose levels.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Groups:
- PF-03084014 in Solid Tumor Participants: PF-03084014 150 mg or 220 mg was administered orally BID to participants with solid tumors as single agent for 21 days per cycle continuously (except for Cycle 1=28 days [with a 7-day washout]). On Cycle 1 Day 1 and Cycle 2 Day 1, only the morning dose was administered. Each participant was to serve as their own control in which PF-03084014 was administered in the morning under either "fed" or "fasted" conditions on Day 1 of Cycle 1 and Cycle 2. The testing order for fed versus fasted conditions was as follows: The first 6 participants in this sub-study were tested under fed followed by fasted conditions, the next 6 participants were tested under fasted followed by fed conditions.
Arm/Group | PF-03084014 in Solid Tumor Participants
Number analyzed (Participants) | 11
ng*hr/mL/mg | 23.71 (115)

30. Secondary Outcome: Dose-normalized AUCtau [AUCtau(dn)] in the Fed State for Solid Tumor Participants
Description: as for outcome 29
Time Frame: as for outcome 25
Population: Solid tumor participants who were enrolled in the food-effect sub-study, started treatment and had evaluable PK data under both fed and fasted states. Due to the limited number of evaluable participants (7 at 150 mg BID and 4 at 220 mg BID for Cmax) and a generally dose-proportional exposure (AUCtau and Cmax), data were combined for 2 dose levels.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-03084014 in Solid Tumor Participants
Number analyzed (Participants) | 11
ng*hr/mL/mg | 22.54 (67)

31. Secondary Outcome: Dose-normalized Cmax [Cmax(dn)] in the Fasted State for Solid Tumor Participants
Description: Cmax(dn) was calculated by maximum observed serum concentration (Cmax) divided by administered dose.
Time Frame: as for outcome 25
Population: Participants who were enrolled in the food-effect sub-study, started treatment and had evaluable PK data under both fed and fasted states. Due to the limited number of evaluable participants (9 at 150 mg BID and 4 at 220 mg BID for Cmax) and a generally dose-proportional exposure (AUCtau and Cmax), data were combined for the 2 dose levels.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-03084014 in Solid Tumor Participants
Number analyzed (Participants) | 13
ng/mL/mg | 6.56 (106)

32. Secondary Outcome: Dose-Normalized Cmax [Cmax(dn)] in the Fed State for Solid Tumor Participants
Description: Cmax(dn) was calculated by maximum observed serum concentration (Cmax) divided by administered dose.
Time Frame: as for outcome 25
Population: Solid tumor participants who were enrolled in the food-effect sub-study, were treated and had evaluable PK data under both fed and fasted states. Due to the limited number of evaluable participants (9 at 150 mg BID and 4 at 220 mg BID for Cmax) and a generally dose-proportional exposure (AUCtau and Cmax), data were combined for the 2 dose levels.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-03084014 in Solid Tumor Participants
Number analyzed (Participants) | 13
ng/mL/mg | 5.22 (64)

33. Secondary Outcome: AUCtau on Cycle 2 Day 1
Description: AUCtau was area under the serum concentration-time profile from time 0 to tau (dosing interval). Data for this outcome measure was planned to be analyzed for two arms only.
Time Frame: Cycle 2 Day 1 (pre-dose and 0.5, 1, 2, 4, 10 and 24 hr post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 8 | 4
ng*hr/mL | 2784 (80) | 11870 (57)

34. Secondary Outcome: Dose-normalized AUCtau [AUCtau (dn)] on Cycle 2 Day 1
Description: AUCtau(dn) was calculated by area under the serum concentration-time profile from time 0 to tau (dosing interval) (AUCtau) divided by administered dose. Data for this outcome measure was planned to be analyzed for two arms only.
Time Frame: Cycle 2 Day 1 (pre-dose and 0.5, 1, 2, 4, 10 and 24 hr post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 8 | 4
ng*hr/mL/mg | 18.6 (80) | 54.0 (57)

35. Secondary Outcome: Cmax on Cycle 2 Day 1
Description: Cmax was the maximum observed serum concentration. Data for this outcome measure was planned to be analyzed for two arms only.
Time Frame: Cycle 2 Day 1 (pre-dose and 0.5, 1, 2, 4, 10 and 24 hr post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 9 | 4
ng/mL | 834.6 (76) | 2640 (63)

36. Secondary Outcome: Dose-normalized Cmax [Cmax (dn)] on Cycle 2 Day 1
Description: Cmax(dn) was calculated by maximum observed serum concentration (Cmax) divided by administered dose. Data for this outcome measure was planned to be analyzed for two arms only.
Time Frame: Cycle 2 Day 1 (pre-dose and 0.5, 1, 2, 4, 10 and 24 hr post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 9 | 4
ng/mL/mg | 5.6 (76) | 12.0 (63)

37. Secondary Outcome: Tmax on Cycle 2 Day 1
Description: Tmax was the time to reach maximum serum concentration (Cmax). Data for this outcome measure was planned to be analyzed for two arms only.
Time Frame: Cycle 2 Day 1 (pre-dose and 0.5, 1, 2, 4, 10 and 24 hr post-dose)
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 9 | 4
hr | 2.00 [1.00 to 4.03] | 1.53 [0.98 to 4.00]

38. Secondary Outcome: Percentage of Solid Tumor Participants With Objective Response (OR)
Description: Objective response (OR) was defined as confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as >=30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study >=4 weeks after initial documentation of response.
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1 and then Day 1 (plus [+] or minus [-] 5 days) of every odd cycle or as clinically indicated, up to Cycle 9; afterwards assessed on Day 1 (+ or -5 days) every 4 cycles
Population: All solid tumor participants who received study treatment, had baseline assessments and at least 1 on study tumor assessment prior to any new anti-cancer therapies were considered evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 18 | 10 | 1
percentage of participants | 33.3 [0.8 to 90.6] | 0 [0.0 to 70.8] | 66.7 [9.4 to 99.2] | 0 [0.0 to 52.2] | 0 [0.0 to 70.8] | 5.6 [0.1 to 27.3] | 10.0 [0.3 to 44.5] | 100 [2.5 to 100.0]

39. Secondary Outcome: Time to Tumor Progression (TTP) for Solid Tumor Participants
Description: Time from Cycle 1 Day 1 to first documentation of disease progression. Progression was defined as per RECIST version 1.0, as a 20% increase in the sum of the longest diameter of target lesions, or target lesions over nadir, uneuivocal progression of non-target disease, or the appearance of new lesions. TTP (months) was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.
Time Frame: Baseline until first documented objective progression (up to maximum of 84 months)
Population: All solid tumor participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 4 | 23 | 16 | 3
months | NA [0.8 to NA] — Data was not estimable due to insufficient number of participants with events. | 1.2 [1.0 to 2.8] | NA [1.7 to NA] — Data was not estimable due to insufficient number of participants with events. | 3.1 [1.0 to NA] — Data was not estimable due to insufficient number of participants with events. | 4.3 [1.6 to 19.5] | 1.6 [1.4 to 6.0] | 1.5 [1.1 to 4.2] | NA [NA to NA] — Data was not estimable due to insufficient number of participants with events.

40. Secondary Outcome: Duration of Response (DR) for Solid Tumor Participants
Description: Time from the first documentation of OR to objective disease progression or death due to any cause. DR was only calculated for participants with an OR. DR (months) was calculated as (date of first documentation of objective progression or death minus date of first documentation of PR or CR plus 1) divided by 30.
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1 and then Day 1 (+ or -5 days) of every odd cycle or as clinically indicated, up to Cycle 9. Afterwards, assessed on Day 1 (+ or -5 days) every 4 cycles (up to maximum of 84 months)
Population: Only solid tumor participants with an OR were analyzed; however, all these participants were censored as of the time of data cut-off on 09 January 2013. Of these 6 participants, 4 participants were still on study with 1 participant discontinued for non-compliance and the other 1 participant missing tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 1
months | NA [NA to NA] — Data was not estimable due to insufficient number of participants with events. | NA [NA to NA] — Data was not estimable due to insufficient number of participants with events. | NA [NA to NA] — Data was not estimable due to insufficient number of participants with events. | NA [NA to NA] — Data was not estimable due to insufficient number of participants with events. | NA [NA to NA] — Data was not estimable due to insufficient number of participants with events.

41. Secondary Outcome: Progression-Free Survival (PFS) for Solid Tumor Participants
Description: PFS was defined as the time from Cycle 1 Day 1 to date of first documentation of progression or death due to any cause. Progression was defined as per RECIST version 1.0, as a 20% increase in the sum of the longest diameter of target lesions, or target lesions over nadir, unequivocal progression of non-target disease, or the appearance of new lesions. PFS (months) was calculated as (the first event date minus the date of first dose of study medication plus 1) divided by 30.
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1 and then Day 1 (+ or - 5 days) of every odd cycle or as clinically indicated, up to Cycle 9; afterwards assessed on Day 1 (+ or -5 days) every 4 cycles (up to maximum of 84 months)
Population: All solid tumor participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 4 | 23 | 16 | 3
months | NA [0.8 to NA] — Unable to calculate as 2 participants were censored and only 1 participant was evaluable. | 1.2 [1.0 to 2.8] | NA [1.7 to NA] — Unable to calculate as 3 participants were censored and only 1 participant was evaluable. | 2.3 [0.4 to NA] — The upper 95% confidence limit can not be determined due to limited number of participants with PFS. | 4.3 [1.6 to 19.5] | 1.6 [1.4 to 6.0] | 1.5 [1.1 to 4.2] | NA [NA to NA] — Unable to calculate as all 3 participants were censored.

42. Secondary Outcome: Percentage of T-ALL/LBL Participants With OR
Description: OR was adapted from International Working Group Response Criteria for Acute Myeloid Leukemia (AML). The response categories of interest were CR, complete response with incomplete hematopoietic recovery (CRi), and PR. CR: ANC >1500/microliter (uL), no circulating blasts. Platelets >100,000/uL, <5% marrow blast cells, no extramedullary disease, bone marrow cellularity >20% with tri-lineage hematopoiesis and <5% marrow blast cells, none of which were neoplastic; CRi: same as CR but ANC may be >1500/uL or platelet count >100,000/uL, no requirement on bone marrow cellularity; PR: same as CR but bone marrow with >= 50% reduction of leukemia blast cells and an absolute blast count between 5% and 25%.
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1 and then Day 1 (+ or - 5 days) of every odd cycle or as clinically indicated, up to Cycle 9 (up to maximum of 84 months)
Population: All T-ALL/LBL participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 8
percentage of participants | 12.5 [0.3 to 52.7]

43. Secondary Outcome: Relapse Free Survival (RFS) for T-ALL/LBL Participants
Description: The RFS of CR was defined as the time from the date of first attaining CR to the date of relapse or death from any cause, whichever occurred first. Similarly, the RFS of CR + CRi (or RFS of CR + CRi + PR) was defined as the time from the date of first attaining CR + CRi (or CR + CRi + PR) to the date of relapse or death from any cause, whichever occurred first.
Time Frame: as for outcome 42
Population: Due to halting of T-AA/LBL participants enrollment and limited number of evaluable participants, data for RFS was not collected.
Arm/Group | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 0

44. Secondary Outcome: Peripheral Blast Count Reduction (PBR) for T-ALL/LBL Participants
Description: PBR was the maximum percentage of peripheral blast count reduction for each participant who received at least one dose of study medication. PBR was derived by the Sponsor from percentage of peripheral blood Blast Count reported by sites.
Time Frame: as for outcome 42
Population: Due to halting of T-AA/LBL participants enrollment and limited number of evaluable participants, data for PBR was not collected.
Arm/Group | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 0

45. Secondary Outcome: Changes in Expression Levels of Notch 1 Target Genes in Tumor Biopsies for Solid Tumor Participants: Hairy and Enhancer of Split-4 (Hes4) Gene Expression Levels on Cycle 1 Day 21 Relative to That at Baseline
Description: Gene expression analysis in tumor biopsies was done using cDNA prepared from RNA extracted from tumor biopsies. Gene expression was measured by custom Taqman low density array (TLDA) cards run on Applied Biosystems 7900HT Fast Real-Time polymerase chain reaction (PCR) system. Changes from baseline were calculated as ratios to baseline. Only Hes4 gene showed consistent down modulation across dosing cohorts (150 mg and 220 mg BID) and therefore results were reported for Hes4 only. Data for this outcome measure was planned to be analyzed for two arms only.
Time Frame: Baseline, Cycle 1 Day 21 (-5 days)
Population: Pharmacodynamic Biomarker analysis set was defined separately for T-ALL and advanced solid tumor malignancy participants. In both cases it will comprise all participants enrolled in study having at least one biomarker assessment at baseline and at least one assessment after being treated. Here, "N" signifies participants evaluable for this OM.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 3 | 2
ratio | 0.9 (0.57) | 0.5 (0.50)

46. Secondary Outcome: Changes From Baseline in Expression Levels of Notch 1 Target Genes in Peripheral Blood for T-ALL/LBL Participants: Hes4 Gene Expression Levels on Cycle 1 Day 8, Cycle 1 Day 15, Cycle 1 Day 21 Relative to That at Baseline
Description: Ribonucleic acid (RNA) was extracted from peripheral blood and used as a template to synthesize complementary deoxyribonucleic acid (cDNA). Gene expression in cDNA was measured by custom Taqman low density array (TLDA) cards run on Applied Biosystems 7900HT Fast Real-Time polymerase chain reaction (PCR) system. Changes from baseline were calculated as ratios to baseline. Results were reported Only for Hes4 as this was the only gene to show consistent down modulation across dosing cohorts (150 mg and 220 mg).
Time Frame: Baseline (morning), Cycle 1 Days 8, 15 and 21 (morning, matched with the first PK sample of the particular day), Cycle 1 Day 21 (24, 48, and 120 hr post-dose) and at end of treatment (EOT)
Population: Pharmacodynamic biomarker analysis set. In both cases, it will comprise all participants enrolled in study having at least 1 biomarker assessment at baseline and at least 1 assessment after being treated. Here, "N"=participants evaluable for this OM. This OM was planned to be analyze for T-ALL/LBL arm only.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 8
ratio
  Cycle 1 Day 8: number analyzed (Participants) | 7
  Cycle 1 Day 8 | 0.7 (0.65)
  Cycle 1 Day 15: number analyzed (Participants) | 4
  Cycle 1 Day 15 | 0.3 (0.41)
  Cycle 1 Day 21: number analyzed (Participants) | 4
  Cycle 1 Day 21 | 0.4 (0.27)
  EOT: number analyzed (Participants) | 1
  EOT | 2.0 (NA) — Data for standard deviation was not estimable since only 1 participant was analyzed.

47. Secondary Outcome: Changes in Expression Levels of Notch 1 Target Genes in Peripheral Blood for Solid Tumor Participants: Hes4 Gene Expression Level on Cycle 1 Day 8 and Cycle 1 Day 21 Relative to That at Baseline
Description: as for outcome 46
Time Frame: Baseline (morning), Cycle 1 Days 8 and 21 (pre-dose)
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 11 | 7
ratio
  Cycle 1 Day 8 | 0.3 (0.24) | 0.1 (0.14)
  Cycle 1 Day 21: number analyzed (Participants) | 6 | 5
  Cycle 1 Day 21 | 0.3 (0.33) | 0.0 (0.02)

48. Secondary Outcome: Changes From Baseline in Notch Intracellular Domain (NICD) Levels in Peripheral Blood for T-ALL/LBL Participants
Description: Notch intracellular domain (NICD) levels was measured in peripheral blood mononuclear cell (PBMC) pellets using a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline, Cycle 1 Days 8 and 15 (pre-dose AM), Cycle 1 Day 21 (pre-dose AM and 24, 48 and 120 hr post-dose) and end of treatment (EOT).
Population: No data were reported for the results of NICD measurement in T-ALL/LBL participants because NICD levels fell below the limit of quantitation of the assay in most cases.
Arm/Group | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 0

49. Secondary Outcome: Changes From Baseline in Notch Intracellular Domain (NICD) Levels in Bone Marrow for T-ALL/LBL Participants
Description: Notch intracellular domain (NICD) was to be measured in bone marrow monoculear cell (BMMC) cell pellets using a validated ELISA.
Time Frame: Baseline, Cycle 1 Day 1 and Cycle 2 Day 1
Population: NICD analyses in bone marrow samples were not done because the number of bone marrow samples received was insufficient and because the analyses were not mandatory per protocol.
Arm/Group | PF-03084014 150 mg BID in T-ALL/LBL Participants
Number analyzed (Participants) | 0

50. Post Hoc Outcome: Time to Response (TTR) for Solid Tumor Participants
Description: Time to response (TTR) was only defined for participants with an objective response (OR). TTR (months) was calculated as (date of first documentation of PR or CR minus date of first dose of study medication plus 1) divided by 30.
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1 and then Day 1 (+ or -5 days) of every odd cycle or as clinically indicated, up to Cycle 9. Afterwards, assessed on Day 1 (+ or -5 days) every 4 cycles.
Population: Only solid tumor participants with an OR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 1
months | 11.2 [NA to NA] — Data for upper and lower limit of 95% CI were not estimable since only 1 participant was analyzed. | 19.4 [8.5 to 30.4] | 2.9 [NA to NA] — Data for upper and lower limit of 95% CI were not estimable since only 1 participant was analyzed. | 10.1 [NA to NA] — Data for upper and lower limit of 95% CI were not estimable since only 1 participant was analyzed. | 5.9 [NA to NA] — Data for upper and lower limit of 95% CI were not estimable since only 1 participant was analyzed.

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (maximum of 84 months)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and non-serious in another participant or 1 participant may have experienced both serious and non-serious event. The safety analysis set includes all enrolled participants who received at least 1 dose of study medication.
Groups:
- PF-03084014 20 mg BID in Solid Tumor Participants: PF-03084014 20 mg was administered orally BID, beginning on Day 1 of each cycle, for 21 days. In Cycle 1 only, participants with advanced solid tumor malignancies received PF-03084014 BID for 21 days (on Cycle 1 Day 21 only the morning dose was administered) followed by 7 days' off-treatment for the purpose of PK assessments. In Cycle 2 and beyond, PF-03084014 was administered BID continuously.
- PF-03084014 150 mg BID in T-ALL/LBL Participants: PF-03084014 150 mg was administered orally BID to participants with T-ALL/LBL as single agent for 21 days per cycle continuously (except for Cycle 1). On Cycle 1 Day 21, only the morning dose was administered, followed by a 7-day washout interval.
Arm/Group | PF-03084014 20 mg BID in Solid Tumor Participants | PF-03084014 40 mg BID in Solid Tumor Participants | PF-03084014 80 mg BID in Solid Tumor Participants | PF-03084014 100 mg BID in Solid Tumor Participants | PF-03084014 130 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in Solid Tumor Participants | PF-03084014 150 mg BID in T-ALL/LBL Participants | PF-03084014 220 mg BID in Solid Tumor Participants | PF-03084014 330 mg BID in Solid Tumor Participants
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 2/4 | 4/8 | 2/4 | 8/23 | 4/8 | 7/16 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 7/8 | 3/4 | 23/23 | 8/8 | 16/16 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PF-03084014 20 mg BID in Solid Tumor Participants (N=3) | PF-03084014 40 mg BID in Solid Tumor Participants (N=3) | PF-03084014 80 mg BID in Solid Tumor Participants (N=4) | PF-03084014 100 mg BID in Solid Tumor Participants (N=8) | PF-03084014 130 mg BID in Solid Tumor Participants (N=4) | PF-03084014 150 mg BID in Solid Tumor Participants (N=23) | PF-03084014 150 mg BID in T-ALL/LBL Participants (N=8) | PF-03084014 220 mg BID in Solid Tumor Participants (N=16) | PF-03084014 330 mg BID in Solid Tumor Participants (N=3)
GRAM POSITIVE COCCI (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1/2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0/2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0/8 | 0 | 0 | 0/2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0/2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0/8 | 0 | 0 | 0/2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 0 | 0/2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/8 | 0 | 0 | 0/2
Disease progression (General disorders) | 0 | 1 | 0 | 1 | 0 | 0/8 | 1 | 2 | 0/2
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0/2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0/8 | 0 | 0 | 0/2
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1/8 | 0 | 0 | 0/2
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0/2
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0/2
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 0 | 0/2
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0/2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0/2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1/2
Arterial injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0/2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 0 | 0/2
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0/2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 1 | 0/2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0/2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0/2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0/2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0/2
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0/2
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0/2
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0/2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2/8 | 0 | 0 | 0/2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 0 | 0/2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1/2
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0/2
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 0 | 0/2
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0/2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0/2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0/2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 0 | 0/2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1/8 | 0 | 0 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PF-03084014 20 mg BID in Solid Tumor Participants (N=3) | PF-03084014 40 mg BID in Solid Tumor Participants (N=3) | PF-03084014 80 mg BID in Solid Tumor Participants (N=4) | PF-03084014 100 mg BID in Solid Tumor Participants (N=8) | PF-03084014 130 mg BID in Solid Tumor Participants (N=4) | PF-03084014 150 mg BID in Solid Tumor Participants (N=23) | PF-03084014 150 mg BID in T-ALL/LBL Participants (N=8) | PF-03084014 220 mg BID in Solid Tumor Participants (N=16) | PF-03084014 330 mg BID in Solid Tumor Participants (N=3)
PRURITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 2/8 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0/8 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Eye movement disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Orbital oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1/8 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2/8 | 1 | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 3/8 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 2/8 | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 3 | 2/8 | 2 | 12 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1/8 | 0 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2/8 | 2 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 1/8 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 3 | 5/8 | 5 | 8 | 2
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2/8 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2 | 5/8 | 5 | 5 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1/8 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0/8 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 1
Early satiety (General disorders) | 1 | 1 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 2 | 1 | 1 | 7/16 | 0 | 7 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Induration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0/8 | 0 | 0 | 1
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 0 | 0 | 2/8 | 0 | 0 | 2
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0 | 0 | 1/8 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 3/8 | 2 | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 1/8 | 0 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1/8 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2/8 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1/8 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0/8 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0/8 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 2/8 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 3/8 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2/8 | 0 | 0 | 0
Urinary tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1/8 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0/8 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0/8 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 1 | 0 | 1/8 | 2 | 0 | 0
Alpha 1 foetoprotein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 1 | 0 | 1/8 | 1 | 2 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0/8 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2 | 1 | 0 | 0/8 | 0 | 0 | 0
Fungal test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Gamma-glutamyltransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0/8 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0/8 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1 | 1 | 7/8 | 0 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 3/8 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1/8 | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 5/8 | 1 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1/8 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 2 | 6/8 | 0 | 9 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 2/8 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 1 | 0 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 1 | 0
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 1
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2/8 | 1 | 0 | 1
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2/8 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 2/8 | 1 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0/8 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0/8 | 2 | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0/8 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0/8 | 0 | 0 | 0
Enuresis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 3/8 | 1 | 3 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Breast disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 0 | 0
Scrotal mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 5/8 | 1 | 5 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 4/8 | 0 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1/8 | 1 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1/8 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 4/8 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1/8 | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0/8 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2/8 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 1 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0/8 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2/8 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2/8 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 0 | 4/8 | 0 | 3 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2/8 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0/8 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1/8 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0/8 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1/8 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1/8 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0/8 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0/8 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study components related to combination therapy with dexamethasone were removed due to operational/scientific reasons. Due to halting of T-AA/LBL participant's enrollment; limited number of evaluable participants, PBR and RFS data was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.